CLINICAL TRIAL: NCT00954772
Title: Mood and STN Deep Brain Stimulation
Brief Title: Mood and Subthalamic Nucleus (STN) Deep Brain Stimulation
Acronym: MOST
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Parkinson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 00056229
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2009-08

CONDITIONS: Movement Disorders
Keywords: Staged versus Simultaneous Bilateral DBS
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Staged Bilateral STN DBS
- Simultaneous Bilateral STN DBS

SUMMARY:
The purpose of this research study is to investigate any changes seen in mood or behavior following deep brain stimulation for movement disorders.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD diagnosed by a movement disorders neurologist
* Approved by a movement disorders neurologist as clinically needing a DBS device
* Absence of significant cognitive dysfunction (Mattis Dementia Rating Scale Score of greater than or equal to 116)
* MRI without evidence of structural abnormality (stroke, tumor, malformation, etc)
* No prior neurosurgical intervention

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients who undergo STN DBS
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2005-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Okun, MD, Principal Investigator — University of Florida
Locations (1):
- Mt. Sinai School of Medicine, New York, New York, United States